CLINICAL TRIAL: NCT01251380
Title: A Phase III, Prospective, Multicentre, Open Label, Extension Study Assessing the Long Term Safety and Efficacy of Repeated Treatment With DYSPORT® Used in the Treatment of Lower Limb Spasticity in Children With Dynamic Equinus Foot Deformity Due to Cerebral Palsy
Brief Title: Dysport® Pediatric Lower Limb Spasticity Follow-on Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-55-52120-147; 2010-019102-17 (EudraCT Number)
Record Dates: First submitted 2010-11-25; First posted 2010-12-01 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy; Muscle Spasticity; Children
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport (Experimental): Dysport was injected into either one or both lower limbs in up to 4 cycles of treatment, a minimum of 12 weeks apart and up to a maximum of 40 weeks apart. Doses varied from 5 Units (U)/Kg to 20 U/kg for one leg, or from 10 U/Kg to 30 U/kg for two legs, with a maximum dose of no more than 30 U/Kg overall, or 1000 U, whichever was reached first.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Intramuscular (IM) injection on day 1 of each treatment cycle.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this research study was to determine the long term safety and efficacy of repeated treatments with Dysport® used in the treatment of lower limb spasticity in children with dynamic equinus foot deformity due to cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for participation in the study if they met the following criteria:

1. Completion of the double blind study (Study 141) up to the Week 12, Week 16, Week 22 or Week 28 follow up visit.
2. Without any major protocol deviations and/or any ongoing adverse events (AEs), either of which, in the opinion of the Investigator would pose an unacceptable risk to the subject were he/she to continue receiving treatment in this open label extension study.
3. Written informed consent obtained from the child's parent(s)/guardian(s) for this study, and assent from the child when and where applicable.

Exclusion Criteria:

Subjects were excluded from entering the study for the following reasons:

1. Major limitation in the passive range of motion at the ankle, as defined by maximum ankle dorsiflexion measured by the angle of arrest (XV1) at slow speed <80° (TS angle) in the most affected leg to be injected.
2. Unwillingness or inability to comply with the protocol.
3. Current need for surgery for spasticity of the gastrocnemius-soleus complex (GSC) and/or hamstring muscles (and/or tendons) in the most affected leg to be injected.
4. Treatment with any drug that interferes either directly or indirectly with neuromuscular function (e.g. aminoglycoside antibiotics) or neuroblocking agents used during surgery (e.g. curare) within the last 30 days prior to study medication or a planned treatment with such drugs.
5. Be pregnant and/or lactating.
6. Female subjects, not willing to use contraceptive measures throughout the course of the study if post pubertal and sexually active.
7. An infection at the injection site(s).
8. Planned treatment with any new investigational drug or device during the study period.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (27):
- United States (8):
  - The Children's Hospital, Aurora, Colorado
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Children's Hospital of Michigan, Detroit, Michigan
  - Gillette Children's Speciality Healthcare, Saint Paul, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriner's Hospital for Children, Portland, Oregon
  - Texas Scottish Rite - Hospital for Children, Dallas, Texas
- Chile (3):
  - Club De Leones Cruz Del Sur Rehabilitation Corporation Punta Arenas, Punta Arenas
  - Dr Roberto Del Rio Hospital, Santiago
  - Neurorehabilitation Laboratory, Pontifical Catholic University, Santiago
- CHU Jean Minjoz, Besançon, France
- Mexico (3):
  - Hospital San José Celaya, Celaya
  - Centro de Rehabilitacion Infantil, Mexico City
  - Centro de Rehabilitacion Integral de Queretaro (CRIQ), Querétaro
- Poland (4):
  - Non-public Healthcare Unit at the Association for Disabled People KROK PO KROKU, Gdansk
  - B i L- Specjalistyczne Centrum Medyczne, Lodz
  - Non-public Healthcare Unit - Grunwaldzka Clinic, Poznan
  - Non-public Healthcare Unit Mazovian Neurorehabilitatio, Wiązowna
- Turkey (Türkiye) (8):
  - Ghulane Military Medical Academy and School of Medicine, Ankara
  - Ibn-i-Sina Hospital, Ankara
  - Yildirim Beyazit Training and Research Hospital, Ankara
  - GATA Haydarpasa Training Hospital, Istanbul
  - Istanbul Fizik Tedavi Rehabilitasyon Egitim ve Arastirma Hastanesi, Istanbul
  - Istanbul University Medical School, Istanbul
  - Dokuz Eylül University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, İzmit

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre study performed at 27 investigational sites in France, Mexico, Turkey, Poland, Chile and the United States of America (USA). Twenty six sites recruited at least one subject and the other site was inactive.
Pre-assignment Details: Of 216 subjects enrolled in this open label study from Study Y-55-52120-141, 203 went straight into Cycle 1. 13 subjects were not considered eligible for re-treatment at end (all of whom had received Dysport) and as per study design they entered into the observational phase of Study 147. Of these 13, 4 subjects entered Cycle 1 at a later date.
Groups:
- Total Dysport: Dysport was injected into the affected GSC with / without Hamstring injections at doses ranging between 5 U/kg to 20 U/kg for one leg and 10 U/kg to 30 U/kg for both legs
Period: Overall Study
Arm/Group | Total Dysport
Started | 216 (Safety population.)
Cycle 1 | 207
Cycle 2 | 175
Cycle 3 | 86
Cycle 4 | 11
Completed | 194
Not Completed | 22
Not completed — Other (Not otherwise specified) | 12
Not completed — Withdrawal by Subject | 6
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Dysport
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (3.3)
Age, Customized [Number; unit: participants]
  Children (2-9 years) | 183
  Children (10-17 years) | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 130
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 5
  Caucasian/White | 159
  American Indian/Alaskan Native | 1
  Multiple | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) Reported in the Double Blind (DB) + Open Label (OL) Period.
Description: Adverse events (AEs) were monitored from the time of informed consent to the end of the study. All AEs were elicited by direct, non-leading questioning or by spontaneous reports.
Time Frame: From baseline (Day 1) until end of study (Week 40) of Cycle 1 and up to Week 28 of Cycles 2 to 4.
Population: Safety Population - all enrolled subjects. One subject received placebo in the DB study and two treatment cycles of Dysport in the OL study. However, as both Dysport treatments were outside of the ranges specified (≤7.5 U/kg in Treatment Cycle 1 and Treatment Cycle 2), the subject was excluded from the analysis (no TEAEs reported for this subject).
Measure: Number; unit: participants
Arm/Group | Total Dysport
Number analyzed (Participants) | 215
participants
  Any TEAE | 177
  Intensity of TEAEs - at least 1 is Severe | 5
  Intensity of TEAEs - at least 1 is Moderate | 91
  Intensity of TEAEs - at least 1 is Mild | 151
  Intensity of TEAEs - at least 1 is Missing | 1
  Causality of TEAEs - at least 1 is Related | 29
  Causality of TEAEs - at least 1 is Not Related | 172
  Causality of TEAEs - at least 1 is Missing | 0
  TEAEs - at least 1 is Related & Severe | 0
  TEAEs - at least 1 is Related & Moderate | 9
  TEAEs - at least 1 is Related & Mild | 23
  TEAEs - at least 1 is Not Related & Severe | 5
  TEAEs - at least 1 is Not Related & Moderate | 87
  TEAEs - at least 1 is Not Related & Mild | 145
  Any TEAEs leading to Study Withdrawal | 1
  Any TEAEs leading to Death | 0
  Any Serious Adverse Events (SAEs) | 7
  Any Non-serious TEAEs | 175

2. Secondary Outcome: Mean Change From Baseline (in the DB Study) in the MAS Score in the GSC Assessed at the Ankle Joint of the (Most) Affected Lower Limb
Description: Baseline for the 'change from DB baseline' was defined as the baseline of Study 141 for all treatment cycles. The Modified Ashworth Scale (MAS) is a 6-point scale which measures the intensity of muscle tone by measuring the resistance of the muscle to passive lengthening or stretching. The investigator graded muscle tone in the GSC from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension).
Time Frame: DB baseline; Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: Intent-to-treat (ITT) population where n represents number of subjects with data. For Dysport 10 U/kg and 15 U/kg, the actual administered doses in the GSC of the (most) affected leg were >7.5 to ≤12.5 U/kg and >12.5 to ≤17.5 U/kg, respectively, in the OL study. The analysis excluded subjects with doses ≤7.5 or >17.5 U/kg.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport
Number analyzed (Participants) | 170
units on a scale
  Treatment Cycle 1, Week 4 (n=170) | -1.0 (0.9)
  Treatment Cycle 1, Week 12 (n=157) | -0.8 (0.8)
  Treatment Cycle 2, Week 4 (n=122) | -1.1 (0.9)
  Treatment Cycle 2, Week 12 (n=93) | -0.9 (0.9)
  Treatment Cycle 3, Week 4 (n=66) | -1.0 (0.8)
  Treatment Cycle 3, Week 12 (n=35) | -0.7 (1.0)
  Treatment Cycle 4, Week 4 (n=8) | -0.4 (0.5)

3. Secondary Outcome: Mean Change From Baseline (Prior to the First Injection Cycle in the Hamstrings) in the MAS Score in the Knee Flexors Assessed at the Knee Joint of the (Most) Affected Lower Limb
Description: Baseline was defined as the value obtained prior to the first injection in the hamstrings. The MAS is a 6-point scale which measures the intensity of muscle tone by measuring the resistance of the muscle to passive lengthening or stretching. The investigator graded muscle tone in the GSC from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension).
Time Frame: Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Baseline and Week 4 of Treatment Cycle 4.
Population: ITT population where n represents number of subjects with data. For Dysport 5 U/kg and 10 U/kg, the actual administered doses in the hamstring of the (most) affected leg were >3 to ≤7.5 U/kg and >7.5 to ≤12.5 U/kg, respectively. Analysis excluded subjects with doses ≤3 or >12.5 U/kg. Only data from subjects injected in the hamstring are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport
Number analyzed (Participants) | 33
units on a scale
  Treatment Cycle 1, Week 4 (n=25) | -0.6 (0.7)
  Treatment Cycle 1, Week 12 (n=24) | -0.8 (0.8)
  Treatment Cycle 2, Week 4 (n=33) | -0.5 (0.9)
  Treatment Cycle 2, Week 12 (n=21) | -0.3 (0.9)
  Treatment Cycle 3, Week 4 (n=13) | -0.2 (0.8)
  Treatment Cycle 3, Week 12 (n=5) | -0.6 (0.5)
  Treatment Cycle 4, Week 4 (n=2) | -0.5 (0.7)

4. Secondary Outcome: Mean Change From Baseline (Prior to the First Injection Cycle in Upper Limb Muscle Groups) in the Mean MAS Score for All Injected Upper Limb Muscle Groups From Treatment Cycle 2 Onwards
Description: Baseline was defined as the value obtained prior to the first injection in the upper limb(s). The MAS is a 6-point scale which measures the intensity of muscle tone by measuring the resistance of the muscle to passive lengthening or stretching. The investigator graded muscle tone in the GSC from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension). No subjects were treated in the upper limb in Treatment Cycle 4.
Time Frame: Baseline and Weeks 4 and 12 of Treatment Cycles 2 and 3.
Population: ITT population where n represents number of subjects with data. Only data from subjects injected in the upper limb muscle groups are presented. TC = Treatment Cycle.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport
Number analyzed (Participants) | 14
units on a scale
  TC 2: Elbow Flexors at Week 4 (n=14) | -1.2 (0.9)
  TC 2: Elbow Flexors at Week 12 (n=12) | -1.1 (0.8)
  TC 2: Wrist Flexors at Week 4 (n=11) | -1.6 (0.8)
  TC 2: Wrist Flexors at Week 12 (n=8) | -1.0 (0.9)
  TC 3: Elbow Flexors at Week 4 (n=2) | 1.0 (0.0)
  TC 3: Elbow Flexors at Week 12 (n=1) | -1.0 (NA) — Non calculable as N=1
  TC 3: Wrist Flexors at Week 4 (n=5) | -1.4 (0.9)
  TC 3: Wrist Flexors at Week 12 (n=2) | -1.5 (0.7)

5. Secondary Outcome: Mean Physician's Global Assessment (PGA) Score
Description: Global assessment of treatment response based on changes since the first injection in the DB study. PGA Scale of the Treatment Response: Global assessment of treatment response was assessed by asking the Investigator the following question: "how would you rate the response to treatment in the subject's lower limb(s) since the first injection in the DB study?" Answers were made on a 9 point rating scale (-4: markedly worse, -3: much worse, -2: worse, -1: slightly worse, 0: no change, +1: slightly improved, +2: improved, +3: much improved, +4: markedly improved).
Time Frame: Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4.
Population: ITT population where n represents number of subjects with data. For Dysport 10 U/kg and 15 U/kg, the actual administered doses in the GSC of the (most) affected leg were >7.5 to ≤12.5 U/kg and >12.5 to ≤17.5 U/kg, respectively. The analysis excluded subjects with doses ≤7.5 or >17.5 U/kg.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport
Number analyzed (Participants) | 195
units on a scale
  Treatment Cycle 1 at Week 4 (n=195) | 1.5 (0.9)
  Treatment Cycle 1 at Week 12 (n=180) | 1.0 (1.2)
  Treatment Cycle 2 at Week 4 (n=159) | 1.5 (1.0)
  Treatment Cycle 2 at Week 12 (n=116) | 0.9 (1.3)
  Treatment Cycle 3 at Week 4 (n=78) | 1.4 (0.9)
  Treatment Cycle 3 at Week 12 (n=37) | 0.7 (1.4)
  Treatment Cycle 4 at Week 4 (n=8) | 0.5 (0.8)

6. Secondary Outcome: Mean Goal Attainment Scale (GAS) Score
Description: Individual goals were defined prior to treatment in each treatment period. The GAS is a functional scale used to measure progress towards individual therapy goals. Individual goals were defined for each subject by the physician, and the child's parents (caregiver) where applicable, prior to treatment. After treatment in each treatment cycle, the GAS for each goal was rated using a defined scale (-2: Much less than expected outcome, -1: Somewhat less than expected outcome, 0: Expected outcome, 1: Somewhat more than expected outcome, and 2: Much more than expected outcome).
Time Frame: Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport
Number analyzed (Participants) | 194
units on a scale
  Treatment Cycle 1 at Week 4 (n=194) | 50.6 (11.0)
  Treatment Cycle 1 at Week 12 (n=178) | 50.7 (10.1)
  Treatment Cycle 2 at Week 4 (n=158) | 51.2 (11.0)
  Treatment Cycle 2 at Week 12 (n=116) | 51.7 (10.5)
  Treatment Cycle 3 at Week 4 (n=78) | 48.3 (10.7)
  Treatment Cycle 3 at Week 12 (n=36) | 45.8 (8.9)
  Treatment Cycle 4 at Week 4 (n=8) | 44.9 (9.4)

7. Secondary Outcome: Mean Change From DB Baseline in Angle of Arrest (XV1) Derived From the Tardieu Scale (TS), in the GSC Assessed at the Ankle Joint of the (Most) Affected Lower Limb
Description: The TS was used to measure spasticity in the GSC at the ankle joint of the (most) affected lower limb.
  The Investigator assessed muscle reactions of the tested muscle to passive stretch at two velocities: SLOW = V1: as slow as possible (slower than the rate of natural drop of the limb segment under gravity); FAST = V2 (speed of the limb segment falling under gravity) or V3 (as fast as possible - faster than the rate of natural drop of the limb segment under gravity).
  The mean change from DB baseline in XV1 at slow speed was derived.
Time Frame: DB baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 169
degrees
  Treatment Cycle 1 at Week 4 (n=169) | 2.6 (9.0)
  Treatment Cycle 1 at Week 12 (n=156) | 1.4 (9.2)
  Treatment Cycle 2 at Week 4 (n=121) | 1.4 (9.2)
  Treatment Cycle 2 at Week 12 (n=92) | 0.4 (10.9)
  Treatment Cycle 3 at Week 4 (n=66) | 0.5 (10.1)
  Treatment Cycle 3 at Week 12 (n=35) | -1.1 (10.4)
  Treatment Cycle 4 at Week 4 (n=8) | -5.0 (9.6)

8. Secondary Outcome: Mean Change From DB Baseline in Angle of Catch (XV3) Derived From the TS, in the GSC Assessed at the Ankle Joint of the (Most) Affected Lower Limb
Description: The TS was used to measure spasticity in the GSC at the ankle joint of the (most) affected lower limb.
  The Investigator assessed muscle reactions of the tested muscle to passive stretch at two velocities: SLOW = V1: as slow as possible (slower than the rate of natural drop of the limb segment under gravity); FAST = V2 (speed of the limb segment falling under gravity) or V3 (as fast as possible - faster than the rate of natural drop of the limb segment under gravity).
  The mean change from DB baseline in XV3 at fast speed was derived.
Time Frame: DB baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Total Dysport: Dysport was injected into the affected GSC with / without Hamstring injections at doses ranging between 5U/kg to 20U/kg for one leg and 10U/kg to 30U/kg for both legs
Arm/Group | Total Dysport
Number analyzed (Participants) | 168
degrees
  Treatment Cycle 1 at Week 4 (n=168) | 12.2 (13.7)
  Treatment Cycle 1 at Week 12 (n=155) | 9.9 (13.7)
  Treatment Cycle 2 at Week 4 (n=119) | 13.3 (12.6)
  Treatment Cycle 2 at Week 12 (n=92) | 11.4 (13.9)
  Treatment Cycle 3 at Week 4 (n=65) | 12.7 (13.4)
  Treatment Cycle 3 at Week 12 (n=35) | 9.9 (14.5)
  Treatment Cycle 4 at Week 4 (n=8) | 4.4 (11.8)

9. Secondary Outcome: Mean Change From DB Baseline in Spasticity Angle (X) Derived From the TS, in the GSC Assessed at the Ankle Joint of the (Most) Affected Lower Limb
Description: The TS was used to measure spasticity in the GSC at the ankle joint of the (most) affected lower limb.
  The Investigator assessed muscle reactions of the tested muscle to passive stretch at two velocities: SLOW = V1: as slow as possible (slower than the rate of natural drop of the limb segment under gravity); FAST = V2 (speed of the limb segment falling under gravity) or V3 (as fast as possible - faster than the rate of natural drop of the limb segment under gravity).
  X (threshold) was derived as XV1 at slow speed minus XV3 at fast speed and the mean change from DB baseline was calculated.
Time Frame: DB Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 168
degrees
  Treatment Cycle 1 at Week 4 (n=168) | -9.7 (12.6)
  Treatment Cycle 1 at Week 12 (n=155) | -8.5 (11.9)
  Treatment Cycle 2 at Week 4 (n=119) | -12.0 (12.0)
  Treatment Cycle 2 at Week 12 (n=92) | -10.9 (12.8)
  Treatment Cycle 3 at Week 4 (n=65) | -12.2 (11.6)
  Treatment Cycle 3 at Week 12 (n=35) | -11.0 (13.4)
  Treatment Cycle 4 at Week 4 (n=8) | -9.4 (8.6)

10. Secondary Outcome: Mean Change From DB Baseline in Spasticity Grade (Y) Derived From the TS, in the GSC Assessed at the Ankle Joint of the (Most) Affected Lower Limb
Description: The mean change from baseline (in the DB study) in Y was derived from the TS.
  Y was graded according to the following scale: Grade 0 - no resistance throughout passive movement (best outcome); Grade 1 - slight resistance throughout passive movement; Grade 2 - clear catch at precise angle, interrupting passive movement, followed by release; Grade 3 - fatigable clonus (less than 10 sec when maintaining pressure) occurring at a precise angle, followed by release; Grade 4 - unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at a precise angle; Grade 5 - joint immovable (worst outcome).
  Catch without release was graded 0 if XV1=XV3, 'unratable' spasticity otherwise; catch with 'minimal' release was graded 2 if XV3 was consistent and consistently less than XV1.
  Angle 0 = position of minimal stretch of the tested muscle. For Grades 0 and 1, spasticity angle X = 0 by definition.
Time Frame: DB Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 169
degrees
  Treatment Cycle 1 at week 4 (n=169) | -0.4 (0.7)
  Treatment Cycle 1 at week 12 (n=155) | -0.3 (0.6)
  Treatment Cycle 2 at week 4 (n=120) | -0.4 (0.7)
  Treatment Cycle 2 at week 12 (n=92) | -0.3 (0.6)
  Treatment Cycle 3 at week 4 (n=66) | -0.4 (0.6)
  Treatment Cycle 3 at week 12 (n=35) | -0.3 (0.6)
  Treatment Cycle 4 at week 4 (n=8) | -0.3 (0.5)

11. Secondary Outcome: Mean Change From Baseline (Prior to the First Injection Cycle in the Hamstrings) in XV1 Derived From the TS, in the Knee Flexors Assessed at the Knee Joint of the (Most) Affected Lower Limb
Description: The TS was used to measure spasticity in the knee flexors at the knee joint of the (most) affected lower limb.
  The Investigator assessed muscle reactions of the tested muscle to passive stretch at two velocities: SLOW = V1: as slow as possible (slower than the rate of natural drop of the limb segment under gravity); FAST = V2 (speed of the limb segment falling under gravity) or V3 (as fast as possible - faster than the rate of natural drop of the limb segment under gravity).
  The mean change from baseline (prior to the first injection cycle in the hamstrings) in XV1 at slow speed was derived.
Time Frame: Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Baseline and Week 4 of Treatment Cycle 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 33
degrees
  Treatment Cycle 1 at Week 4 (n=26) | 3.2 (10.0)
  Treatment Cycle 1 at Week 12 (n=24) | 6.9 (10.4)
  Treatment Cycle 2 at Week 4 (n=33) | 3.0 (11.4)
  Treatment Cycle 2 at Week 12 (n=21) | 5.5 (11.4)
  Treatment Cycle 3 at Week 4 (n=13) | 3.8 (12.1)
  Treatment Cycle 3 at Week 12 (n=5) | 2.0 (7.6)
  Treatment Cycle 4 at Week 4 (n=2) | 5.0 (7.1)

12. Secondary Outcome: Mean Change From Baseline (Prior to the First Injection Cycle in the Hamstrings) in XV3 Derived From the TS, in the Knee Flexors Assessed at the Knee Joint of the (Most) Affected Lower Limb
Description: The TS was used to measure spasticity in the knee flexors at the knee joint of the (most) affected lower limb.
  The Investigator assessed muscle reactions of the tested muscle to passive stretch at two velocities: SLOW = V1: as slow as possible (slower than the rate of natural drop of the limb segment under gravity); FAST = V2 (speed of the limb segment falling under gravity) or V3 (as fast as possible - faster than the rate of natural drop of the limb segment under gravity).
  The mean change from baseline (prior to the first injection cycle in the hamstrings) in XV3 at fast speed was derived.
Time Frame: Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Baseline and Week 4 of Treatment Cycle 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 33
degrees
  Treatment Cycle 1 at Week 4 (n=26) | 10.1 (14.8)
  Treatment Cycle 1 at Week 12 (n=24) | 13.3 (16.3)
  Treatment Cycle 2 at Week 4 (n=33) | 8.2 (15.1)
  Treatment Cycle 2 at Week 12 (n=21) | 12.4 (16.5)
  Treatment Cycle 3 at Week 4 (n=13) | 11.9 (22.3)
  Treatment Cycle 3 at Week 12 (n=5) | 30.0 (24.5)
  Treatment Cycle 4 at Week 4 (n=2) | 5.0 (7.1)

13. Secondary Outcome: Mean Change From Baseline (Prior to the First Injection Cycle in the Hamstrings) in X Derived From the TS, in the Knee Flexors Assessed at the Knee Joint of the (Most) Affected Lower Limb
Description: The TS was used to measure spasticity in the knee flexors at the knee joint of the (most) affected lower limb.
  The Investigator assessed muscle reactions of the tested muscle to passive stretch at two velocities: SLOW = V1: as slow as possible (slower than the rate of natural drop of the limb segment under gravity); FAST = V2 (speed of the limb segment falling under gravity) or V3 (as fast as possible - faster than the rate of natural drop of the limb segment under gravity).
  X (threshold) was derived as XV1 at slow speed minus XV3 at fast speed and the mean change from baseline (prior to the first injection cycle in the hamstrings) was calculated.
Time Frame: Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Baseline and Week 4 of Treatment Cycle 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 33
degrees
  Treatment Cycle 1 at Week 4 (n=26) | -6.9 (11.3)
  Treatment Cycle 1 at Week 12 (n=24) | -6.5 (11.8)
  Treatment Cycle 2 at Week 4 (n=33) | -5.2 (12.0)
  Treatment Cycle 2 at Week 12 (n=21) | -6.9 (11.8)
  Treatment Cycle 3 at Week 4 (n=13) | -8.1 (13.6)
  Treatment Cycle 3 at Week 12 (n=5) | -28.0 (20.8)
  Treatment Cycle 4 at Week 4 (n=2) | 0.0 (14.1)

14. Secondary Outcome: Mean Change From Baseline (Prior to the First Injection Cycle in the Hamstrings) in Y Derived From the TS, in the Knee Flexors Assessed at the Knee Joint of the (Most) Affected Lower Limb
Description: The mean change from baseline (prior to the first injection cycle in the hamstrings) in Y was derived from the TS.
  Y was graded according to the following scale: Grade 0 - no resistance throughout passive movement (best outcome); Grade 1 - slight resistance throughout passive movement; Grade 2 - clear catch at precise angle, interrupting passive movement, followed by release; Grade 3 - fatigable clonus (less than 10 sec when maintaining pressure) occurring at a precise angle, followed by release; Grade 4 - unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at a precise angle; Grade 5 - joint immovable (worst outcome).
  Catch without release was graded 0 if XV1=XV3, 'unratable' spasticity otherwise; catch with 'minimal' release was graded 2 if XV3 was consistent and consistently less than XV1.
  Angle 0 = position of minimal stretch of the tested muscle. For Grades 0 and 1, spasticity angle X = 0 by definition.
Time Frame: Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Baseline and Week 4 of Treatment Cycle 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Dysport
Number analyzed (Participants) | 33
degrees
  Treatment Cycle 1 at Week 4 (n=26) | -0.1 (0.6)
  Treatment Cycle 1 at Week 12 (n=24) | -0.1 (0.5)
  Treatment Cycle 2 at Week 4 (n=33) | 0.0 (0.6)
  Treatment Cycle 2 at Week 12 (n=21) | -0.1 (0.6)
  Treatment Cycle 3 at Week 4 (n=13) | -0.1 (0.3)
  Treatment Cycle 3 at Week 12 (n=5) | -0.4 (0.9)
  Treatment Cycle 4 at Week 4 (n=2) | 0.0 (0.0)

15. Secondary Outcome: Mean Change From DB Baseline in the Observational Gait Scale (OGS) Total Score of the (Most) Affected Leg
Description: The OGS is a measurement tool used to objectively quantify positive and negative features (impairments) of the upper motor neurone syndrome. The OGS is useful when children are too young or insufficiently cooperative for instrumented gait analysis. It is based on the Physicians Rating Scale but has some modifications to improve its sensitivity to detect changes following administration of Botulinum Toxin Type A (BTX-A).
  The OGS total score was calculated as the sum of the individual question scores for Questions 1 to 7, with the highest possible score being 20. The parameters collected were: knee position in midstance, initial foot contact, foot contact at midstance, timing of heel raise, hindfoot at midstance, base of support and gait assistive devices. Higher scores indicate better gait.
  The mean change from baseline (in the DB study) in the OGS total score of the (most) affected leg was derived.
Time Frame: DB Baseline and Weeks 4 and 12 of Treatment Cycles 1 to 3; Week 4 of Treatment Cycle 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport
Number analyzed (Participants) | 178
units on a scale
  Treatment Cycle 1 at Week 4 (n=178) | 1.0 (3.0)
  Treatment Cycle 1 at Week 12 (n=166) | 0.3 (2.8)
  Treatment Cycle 2 at Week 4 (n=142) | 1.4 (3.0)
  Treatment Cycle 2 at Week 12 (n=104) | 0.8 (2.8)
  Treatment Cycle 3 at Week 4 (n=70) | 1.4 (3.2)
  Treatment Cycle 3 at Week 12 (n=35) | 1.0 (2.6)
  Treatment Cycle 4 at Week 4 (n=8) | 0.3 (3.8)

16. Secondary Outcome: Mean Change From DB Baseline in the PedsQL Score (CP Module Scores) at Each Study Visit Except Week 4
Description: The PedsQL has a disease specific CP module that is relevant to the study population and complements the core modules.
  The 35-item questionnaire encompassed 7 scales including (1) daily activities (2) school activities (3) movement and balance (4) pain and hurt (5) fatigue (6) eating activities and (7) speech and communication. A 5-point scale was utilised for parent proxy-report: 0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem.
  Each CP score was calculated as follows: (1) Individual item scores were reversed and transformed from a 0-4 scale to a 0-100 scale by assigning 0=100, 1=75, 2=50, 3=25 and 4=0; (2) Each scale score was calculated as the sum of the transformed individual item scores, divided by the number of non-missing items. Higher scores indicated better quality of life (fewer symptoms or problems).
  A scale score was only calculated if at least 50% of the associated items were non-missing.
Time Frame: Baseline and Week 12
Population: ITT population where n represents number of subjects with data. For Treatment Cycle 4, Week 12 was not included in the study design. Subjects who completed the study or withdrew were counted as missing at subsequent visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dysport Treatment Cycle 1; Dysport Treatment Cycle 2; Dysport Treatment Cycle 3: Dysport was injected into the affected GSC with / without Hamstring injections at doses ranging between 5 U/kg to 20 U/kg for one leg and 10 U/kg to 30 U/kg for both legs
Arm/Group | Dysport Treatment Cycle 1 | Dysport Treatment Cycle 2 | Dysport Treatment Cycle 3
Number analyzed (Participants) | 179 | 120 | 39
units on a scale
  Daily activities at Week 12 (n=178, n=119, n=39) | 6.9 (18.6) | 9.2 (20.8) | 14.4 (19.0)
  Movement and balance at Week 12 (n=179,n=120,n=39) | 7.7 (21.0) | 8.9 (19.6) | 13.5 (19.3)
  Fatigue at Week 12 (n=178, n=120, n=39) | 4.7 (19.0) | 5.0 (18.4) | 9.0 (17.0)
  Pain and hurt at Week 12 (n=179, n=120, n=39) | 3.5 (17.9) | 4.5 (16.2) | 2.7 (21.3)
  School activities at Week 12 (n=103, n=71, n=26) | 3.8 (24.5) | 5.1 (20.4) | 7.7 (14.5)
  Eating activities at Week 12 (n=178, n=120, n=39) | 2.0 (15.2) | 2.1 (14.9) | 2.7 (10.8)
  Speech&Communication at week 12(n=103, n=72, n=26) | 2.5 (17.4) | 2.3 (16.1) | 5.8 (16.5)

17. Secondary Outcome: Mean Change From DB Baseline in the PedsQL Score (Generic Core Scores) at Each Study Visit Except Week 4
Description: The PedsQL is a validated quality of life questionnaire, designed for children from 2 to 18 years of age. The Generic Core Scale covers four multidimensional scales including physical, emotional, social and school aspects, with three summary scales of total scale score, physical health summary score and psychosocial health summary score.
  Each generic core scale was calculated as follows: (1) Individual item scores were reversed and transformed from a 0-4 scale to a 0-100 scale by assigning 0=100, 1=75, 2=50, 3=25 and 4=0; (2) Each scale score was calculated as the sum of the transformed individual item scores, divided by the number of non-missing items. Higher scores indicated better quality of life (fewer symptoms or problems).
  A scale score was only calculated if at least 50% of the associated items were non-missing.
Time Frame: Baseline and Week 12
Population: ITT population where n represents number of subjects with data. For Treatment Cycle 4, Week 12 was not included in the study design. Subjects who completed the study or withdrew were counted as missing at subsequent visits. PHS = pyschosocial health summary; W12 = Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Treatment Cycle 1 | Dysport Treatment Cycle 2 | Dysport Treatment Cycle 3
Number analyzed (Participants) | 174 | 119 | 39
units on a scale
  Physical health summary (W12) (n=173, n=119, n=39) | 7.8 (17.2) | 6.1 (20.9) | 8.0 (20.6)
  PHS (W12) (n=174, n=118, n=39) | 4.1 (13.5) | 4.6 (13.8) | 8.9 (12.1)
  Total Scale (W12) (n=173, n=119, n=39) | 5.5 (12.5) | 5.2 (13.9) | 8.6 (13.6)

ADVERSE EVENTS:
Time Frame: From Day 1 to end of study (week 40)
Description: Safety population. One subject received placebo in the DB study and two cycles of Dysport in the OL study. As both Dysport treatments were outside of the ranges specified (≤7.5 U/kg in Treatment Cycles 1 and 2), the subject was excluded from the analysis (no TEAEs were reported for this subject), and the number of participants at risk was equal to 215.
  A total of 175 subjects experienced nonserious AEs, of whom 147 experienced nonserious AEs that occurred above the frequency threshold of 5%.
Arm/Group | Total Dysport
Serious Adverse Events (participants affected / at risk) | 7/215
Other Adverse Events (participants affected / at risk) | 147/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport (N=215)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (2)
Complex Partial Seizures (Nervous system disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport (N=215)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24)
Pyrexia (General disorders) | 34 (43)
Diarrhoea (Gastrointestinal disorders) | 16 (18)
Vomiting (Gastrointestinal disorders) | 12 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (13)
Upper Respiratory Tract Infection (Infections and infestations) | 46 (71)
Nasopharyngitis (Infections and infestations) | 47 (65)
Influenza (Infections and infestations) | 20 (28)
Pharyngitis (Infections and infestations) | 25 (32)
Bronchitis (Infections and infestations) | 19 (23)
Varicella (Infections and infestations) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A plan for scientific publication and presentation of the results could be agreed and implemented by the study investigators or a steering committee. The sponsor required that reasonable opportunity be given to review the content and conclusions of any abstract, presentation, or paper before the material was submitted for publication or communicated. This condition also applied to any amendments that were subsequently requested by referees or journal editors.